CLINICAL TRIAL: NCT06321198
Title: A Trial to Evaluate the Safety and Preliminary Efficacy of Human Induced Pluripotent Stem Cell Derived Mesenchymal Stromal Cells in Subjects With Steroid-refractory Acute Graft-Versus-Host Disease
Brief Title: A Trial to Evaluate the Safety and Preliminary Efficacy of iMesenchymal Stromal Cells(iMSC) in Subjects With SR-aGVHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xiaoyu Zhu, Chief physician, Anhui Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iMSC-2001
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Steroid-refractory Acute Graft-versus-host Disease(SR-aGVHD)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iMSC injection (Experimental): Low dose injection once a week; Low dose injection twice a week; High dose injection once a week; High dose injection twice a week;
  Interventions: Biological: iMSC

INTERVENTIONS:
Biological: iMSC — Subjects will receive 4 or more times of iMSC injection

SUMMARY:
A study to evaluate the safety and preliminary efficacy of iMSC in subjects with SR-aGVHD

DETAILED DESCRIPTION:
A single center, open label, dose escalation study to evaluate the safety,tolerability and preliminary efficacy of iMSC in subjects with SR-aGVHD

ELIGIBILITY:
Inclusion Criteria:

1.Subjects who understand and voluntarily sign the Informed Consent Form(ICF); 2.4-70 years; 3.Subjects with SR-aGVHD; 4.ECOG≤2; 5.Subjects with II to IV grades of steroid hormone resistance;

Exclusion Criteria:

1. Accepted systemic or local treatment of mesenchymal stem cells;
2. Have severe allergy to blood products or have allergy history of heterologous protein;
3. Expected survival period within 3 months;
4. Alanine transaminase(ALT)or Aspartate aminotransferase(AST)>2*upper limit of normal(ULN);Creatinine clearance rate≤30ml/min or Blood Urea Nitrogen(BUN)>2*upper limit of normal(ULN), International Normalized Ratio (INR)>1.5*upper limit of normal(ULN);
5. Have severe hepatic veno-occlusive disease(HVOD);
6. Have severe lung disease like severe lung infection;
7. Have history of severe acute myocardial infarction or have uncontrolled angina pectoris,arrhythmia and severe heart failure;
8. Proved having resistant hypertension within 6 months before enrollment;
9. Have active thrombus;
10. Have untreated or uncertain active solid tumors within 5 years;
11. Have alcohol or drug addiction or with a clear history of mental disorders or with a history of drug abuse or drug use of psychotropic substances;
12. Human immunodeficiency virus(HIV)antibody positive, treponema pallidum (TP) antibody positive;
13. Have active hepatitis B or hepatitis C;
14. Have gastrointestinal symptoms which not caused by GVHD
15. Pregnant or lactating female subjects, or subjects who are unable to comply with contraceptives from the study period to 6 months after the end of this study;
16. Subjects who have participated in other clinical trials and have used other study products within 12 weeks before screening;
17. Not suitable for this clinical trial for other reasons.

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-02-10 (Actual); Primary Completion 2027-03-02 (Estimated); Study Completion 2027-03-02 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity(DLT) | 4 weeks after initial infusion
  Number of Dose-limiting toxicity in 28 days after injection
Adverse Event(AE),Serious Adverse Event(SAE),Treatment Emergent Adverse Event(TEAE)and Treatment Related Adverse Event(TRAE) | From the date of initial infusion to 180 days after initial infusion
  Number of treatment-related adverse events,treatment emergent adverse event,treatment related adverse event or serious adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | 28 days after initial infusion
  Percentage of participants achieved Complete Response(CR) or Partial Response(PR)
Overall Survival(OS) | 100 days after initial infusion
  The time from initial infusion to death

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Zhu, PH.D, Principal Investigator — Anhui Provincial Hospital
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China